CLINICAL TRIAL: NCT06365606
Title: A Prospective Cross-Sectional Study to Evaluate Diagnostic Sensitivity and Specificity of iStatis Syphilis Ab Test at the Point- Of-Care Sites
Brief Title: Study to Evaluate Diagnostic Sensitivity and Specificity of iStatis Syphilis Ab Test at the Point- Of-Care Sites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: bioLytical Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: CLS-015A
Record Dates: First submitted 2024-04-09; First posted 2024-04-15 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Syphilis Infection; Syphilis
Keywords: syphilis rapid test; syphilis point of care tests; syphilis antibody test; iStatis Syphilis Ab Test; iStatis Syphilis Antibody Test
MeSH Terms: conditions — Syphilis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participants and the healthcare providers are not aware of the syphilis status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Performance onsite (Experimental): Capillary (fingerstick) blood samples collected from the participants will be tested with the iStatis Syphilis Ab Test in the hands of trained healthcare professionals at the point-of-care setting.
  Interventions: Device: iStatis Syphilis Ab Test
- Performance in lab (Experimental): Venous whole blood and plasma samples collected from the participants will be tested with the iStatis Syphilis Ab Test in the hands of trained healthcare professionals at the point-of-care setting. The results are compared with Abbott Architect Syphilis Tp (EDA) referent test, and in cases of positive results, further confirmatory testing (BD Macro-Vue Particle Agglutination (RPR) and Serodia Particle Agglutination (TPPA)) will be conducted.
  Interventions: Device: iStatis Syphilis Ab Test

INTERVENTIONS:
Device: iStatis Syphilis Ab Test — Capillary (fingerstick) blood, venous whole blood and plasma samples prospectively collected from the participants will be tested on the iStatis Syphilis Ab Test.

SUMMARY:
This study is a prospective cross-sectional study in which surgically non-invasive sample- taking is done only for the purpose of the study. Capillary (fingerstick) whole blood and plasma (i.e., obtained through venous EDTA whole blood collection and processing) are collected by a healthcare professional. The collected samples are tested in a routine testing environment, i.e., healthcare providers at

DETAILED DESCRIPTION:
A trained healthcare provide will collect 50μL of capillary whole blood and 11mL of EDTA venous whole blood (VWB) to be tested with the iStatis Syphilis Ab Test on site according to the 'Test Procedure' described in the Instructions for Use (IFU) supplied with the reagents. Same procedure must be followed using the extracted plasma sample to test 30μL of the plasma sample extracted and obtained through processing of the VWB on the iStatis Syphilis Ab Test. An aliquot of the plasma sample will be transferred to the central laboratory to establish the reference test result using an enzyme immunoassay (EIA) (Abbott Architect Syphilis Tp EDA). In case of positive results in the EIA reference test of (Abbott Architect Syphilis Tp EDA), the sample will be sent for BD Macro-Vue Particle Agglutination (RPR) and Serodia Particle Agglutination (TPPA) testing.

ELIGIBILITY:
Inclusion Criteria:

* Participants/subjects (males, females, and pregnant women) getting tested for syphilis for one or more of the following reasons:

  o at risk for syphilis ohaving signs and symptoms indicative for syphilis oRoutine testing
* Participants/subjects of 18 years or older and, who are able to give/sign the informed consent.

Exclusion Criteria:

* Participant younger than 18 years old
* Participants unable to provide written informed consent
* Participants currently undergoing treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2024-03-14 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of the iStatis Syphilis Ab Test | 15 weeks
  To evaluate the diagnostic sensitivity and diagnostic specificity of the iStatis Syphilis Antibody Test at Point-Of-Care (POC).

CONTACTS AND LOCATIONS:
Locations (1):
- Epicentre Health Research, Hillcrest, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: No